CLINICAL TRIAL: NCT01883011
Title: Randomized, Double Blind, Placebo Controlled, Two Parallel Group Study to Evaluate the Efficacy and Safety of Piracetam, 12 g Intravenous (IV) Infusion Within 7 Hour (h) Post Stroke Onset, Followed by 12 g/d for 4 Weeks (IV Ampoules, Oral Solution) and 4.8 g/d for 8 Weeks (Tablets) in Adult Subjects With an Acute Ischemic Middle Cerebral Artery Stroke
Brief Title: A Study to Evaluate the Efficacy and Safety of Piracetam on Aphasia After Acute Ischemic Cerebral Artery Stroke
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated after a pre-specified interim analysis. Please see Detailed Study Description for further information.
Sponsor: UCB S.A. - Pharma Sector (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N09642
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Acute Ischaemic Middle Cerebral Artery Stroke
Keywords: Piracetam; Stroke; Aphasia; Acute; Cerebral; Ischemic; Nootropil
MeSH Terms: conditions — Stroke; Aphasia; Ischemia | interventions — Piracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piracetam (Experimental): IV infusion 12 g piracetam in 60 ml
  IV Ampoules 3 g piracetam in 15 ml
  Oral solution 33 % piracetam (bottle of 125 ml)
  Oral tablets 1200 mg piracetam (blisters of 10 tablets)
  Interventions: Drug: Piracetam
- Placebo (Placebo Comparator): IV infusion 12 g placebo in 60 ml
  IV Ampoules 3 g placebo in 15 ml
  Oral solution 33% placebo (bottle of 125 ml)
  Oral tablets 1200 mg placebo (blisters of 10 tablets)
  All IV forms were identical in presentation, size and color to allow a double blind design.
  All oral forms were identical in shape, size, color and taste to allow a double blind design.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Piracetam
  Arms: Piracetam
Other: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study was to confirm the efficacy of piracetam after 12 weeks of treatment on the aphasic status of subjects suffering from aphasia after acute ischemic middle cerebral artery stroke and having received their medication within 7 h post-stroke onset.

DETAILED DESCRIPTION:
An interim analysis was performed, as planned in the protocol, on the primary efficacy measure (Day 84 FAST Score) for aphasic subjects. This interim analysis indicated that there was less than a 20 % chance of showing a 15 % difference between placebo and piracetam at the end of the trial, under the assumption that there was indeed a 15 % difference. Thus, it was the decision of UCB to stop further recruitment into this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 50 years
* Considered as reliable and mentally capable of adhering to the protocol
* Signed informed consent (by the subject or the next of kin) or inclusion of the subject as per Ethics Committee approved procedures
* Clinical diagnosis of a middle cerebral artery ischemic stroke
* A disabling motor deficit at the moment of inclusion, defined as having a total Middle Cerebral Artery (MCA) score between 15 and 65
* Treated before 7 h (6 h and 59 minutes) after the estimated stroke onset
* If the subject had a stroke during the night, the onset of stroke is assumed to be the last time the subject was seen awake and normal, or last time the subject remembered he/she was awake and normal
* Being aphasic, defined as having an Aphasia Severity Rating (ASR) score of < 3

Exclusion Criteria:

* Stupor or coma: < 10 on the item consciousness of the Middle Cerebral Artery (MCA) scale
* A previous stroke with clinical sequel or a previous stroke with aphasia (even in case of complete recovery from aphasia)
* A medical or neurological disease interfering with the assessments and causing a clear deficit:
* 1. in functional ability or autonomy
* 2. in motor function
* 3. in cognitive capacities
* 4. in language
* A systemic disease with neurological symptoms
* A life threatening disease with life expectancy of less than 1 year
* Renal insufficiency (creatinine > 2 mg/100 ml or > 180 µmol/l; creatinine had to be determined as soon as possible but not before inclusion)
* Any concomitant treatments that could not be stopped at the moment of inclusion or that had been started after the onset of the stroke and before inclusion (as long as not considered by the advisory board as effective drug), such as:
* 1. Cerebro-vascular active products: bufenine, buflomedil, cinnarizine, codergocrinemesilate, citicholine, cyclandelate, cyprodemanol, deanolacetamidobenzoate, flunarizine, ginkgo-biloba extr., inositolnicotinate, isoxsuprine, meclofenoxate, naftidrofuryloxalate, nicergoline, nicotinic acid (smoking is allowed), nimodipine, pentifylline, papaverine, pentoxifylline, piracetam, pyrisuccideanoldimaleate, pyritinol, raubasine, vincamine, viquidil, xantinolnicotinate. A list of these drugs with generic and brand name, adapted to each of the participating countries accompanied the Case Report Form (CRF)
* 2. Thrombolytics: recombinant tissue-type plasminogen activator (alteplase) (rt- PA), streptokinase, urokinase, ancrod
* 3. Hemodilution
* 4. Glucose infusion >5 %
* Subjects known to not being able to be followed for 12 weeks
* Known alcohol or drug addiction or abuse
* Subjects previously enrolled in this trial
* Known allergy/intolerance to piracetam/excipients
* Lactation, pregnancy, or pregnancy potential, unless using an effective means of contraception
* Illiterate subjects (subjects not able to read prior to stroke)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 1998-08; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects recovering from aphasia as per the Frenchay Aphasia Screening Test (FAST) score at Day 84 | Day 84
  FAST describes the presence, absence or severity of aphasia, but does not differentiate types of aphasia.
  Comprehension, expression and reading were main score targets tested by picture card with attached reading card. The FAST score covered a range from 0-20. Subjects with FAST score ≤13 where considered as aphasic and subjects with FAST score > 13 were considered as non-aphasic.
  There were 2 tests of comprehension and 2 tests of expression and 1 of reading, however the reading test was not included in the primary efficacy variable.

SECONDARY OUTCOMES:
Middle Cerebral Artery infarction scale (MCA) score at Day 84 | Day 84
  The MCA was developed for clinical trial evaluation of middle cerebral artery stroke. The scale evaluates 10 items: consciousness, verbal communication, elevation of the arm, finger and thumb movements, arm tone, deviation of head and eyes, facial movements, elevation of the leg, dorsiflexion of the foot and leg tone. Weighted scores for each item provide a maximum score of 100.
Total Barthel Index (BI) score at Day 84 | Day 84
  This scale evaluates 10 items: eating, moving from (wheel) chair to bed and back, personal hygiene, using the lavatory, bathing, walking/wheelchair, stairs, getting dressed/undressed, controlling bowel motion, controlling bladder.
  Weighted scores for each item vary between 0 and 15 to provide a maximum score of 100. Subjects who can perform all specified activities without help receive a score of 100. Even though they are independent in daily activities, they could remain handicapped by neurologic impairments.
Mini Mental State Examination (MMSE) score at Day 84 | Day 84
  The MMSE is divided into two sections, the first of which requires vocal responses only and covers orientation, memory and attention: the maximum score is 21.
  The second part tests ability to name, follow verbal and written commands, write a sentence spontaneously and copy a complex polygon: the maximum score is 9. Maximum score of the two parts is 30. The test is not timed. A score ≤ 23 indicates that the subject is demented.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (44):
- Argentina (2):
  - 050, Buenos Aires
  - 051, Buenos Aires
- Austria (3):
  - 004, Inssbruck
  - 001, Linz
  - 003, Linz
- Belgium (4):
  - 102, Antwerp
  - 103, Antwerp
  - 104, Brussels
  - 107, Genk
- France (2):
  - 150, Charleville-Mézières
  - 152, Nice
- Germany (4):
  - 201, Magdeburg
  - 200, Minden
  - 203, Nidda-bad-Salzhausen
  - 202, Saarbrücken
- Greece (6):
  - 251, Athens
  - 252, Athens
  - 302, Budapest
  - 303, Budapest
  - 305, Budapest
  - 250, Thessaloniki
- Hungary (3):
  - 300, Budapest
  - 304, Debrecen
  - 301, Miskolc
- 350, Perugia, Italy
- 750, Bergen, Norway
- Poland (6):
  - 455, Bialystok
  - 454, Krakow
  - 456, Lodz
  - 451, Poznan
  - 450, Warsaw
  - 452, Warsaw
- Singapore (2):
  - 600, Singapore
  - 601, Singapore
- Spain (4):
  - 501, Madrid
  - 502, Madrid
  - 503, Málaga
  - 500, Terrassa
- 550, Stockholm, Sweden
- 700, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - 654, Edirne
  - 650, Eskişehir
  - 652, Istanbul
  - 653, Istanbul